CLINICAL TRIAL: NCT02964013
Title: A Phase 1 Trial of MK-7684 as Monotherapy and in Combination With Pembrolizumab in Subjects With Advanced Solid Tumors
Brief Title: Study of Vibostolimab Alone and in Combination With Pembrolizumab in Advanced Solid Tumors (MK-7684-001) ( KEYVIBE-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7684-001; MK-7684-001 (Other: Merck); 194809 (Registry Identifier: JAPAC-CTI); KEYVIBE-001 (Other: Merck)
Record Dates: First submitted 2016-11-11; First posted 2016-11-15 (Estimated); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Neoplasms
Keywords: Programmed Cell Death Receptor 1 (PD-1); Programmed Cell Death Receptor Ligand 1 (PD-L1); Programmed Cell Death Receptor Ligand 2 (PD-L2); PD-1; PDL1; PD-L1; PD-L2
MeSH Terms: conditions — Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Pemetrexed; Carboplatin; Cisplatin; Etoposide; etoposide phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- vibostolimab (Experimental): During an initial dose evaluation phase, participants will receive Dose A, B, C, D, E, or F of vibostolimab on Day 1 of each 21-day infusion cycle (for a maximum of 35 cycles) until the RPTD has been established. The RPTD will be established based on the number of dose limiting toxicities (DLTs) at each dose level. Once the RPTD is established, participants will continue receiving the RPTD of vibostolimab on Day 1 of each 21-day infusion cycle until the 35-cycle limit is reached.
  Interventions: Biological: vibostolimab
- vibostolimab + pembrolizumab (Experimental): During an initial dose evaluation phase, participants will receive Dose A, B, C, D, E, or F of vibostolimab in combination with 200 mg pembrolizumab on Day 1 of each 21-day infusion cycle (for a maximum of 35 cycles) until the RPTD of vibostolimab has been established. The RPTD will be established based on the number of DLTs at each dose level. Once the RPTD of vibostolimab is established, participants will continue receiving the RPTD of vibostolimab in combination with 200 mg pembrolizumab on Day 1 of each 21-day infusion cycle until the 35-cycle limit is reached.
  Interventions: Biological: vibostolimab; Biological: pembrolizumab
- Advanced solid tumor cohort (Experimental): Participants will receive the RPTD of vibostolimab monotherapy or the RPTD of vibostolimab in combination with 200 mg pembrolizumab on Day 1 of each 21-day infusion cycle until the 35-cycle limit is reached.
  Interventions: Biological: vibostolimab; Biological: pembrolizumab
- Randomized dose 1 comparison cohort (Experimental): Participants will be randomized to receive a fixed dose (Dose 1) of vibostolimab in combination with 200 mg pembrolizumab on Day 1 of each 21-day infusion cycle until the 35-cycle limit is reached.
  Interventions: Biological: vibostolimab; Biological: pembrolizumab
- Randomized dose 2 comparison cohort (Experimental): Participants will be randomized to receive a fixed dose (Dose 2) of vibostolimab in combination with 200 mg pembrolizumab on Day 1 of each 21-day infusion cycle until the 35-cycle limit is reached.
  Interventions: Biological: vibostolimab; Biological: pembrolizumab
- vibostolimab +pembrolizumab+pemetrexed+carboplatin (Experimental): Participants will receive a fixed dose of vibostolimab in combination with 200 mg pembrolizumab, 500 mg/m^2 pemetrexed, and Area Under Curve (AUC) 5 mg/mL/min carboplatin on Day 1 of each 21-day infusion cycle for up to 4 cycles followed by maintenance therapy with a fixed dose of vibostolimab in combination with 200 mg pembrolizumab and 500 mg/m^2 pemetrexed on Day 1 of each 21-day infusion cycle for up to an additional 31 cycles.
  Interventions: Biological: vibostolimab; Biological: pembrolizumab; Drug: pemetrexed; Drug: carboplatin
- vibostolimab Dose 1 Japanese cohort (Experimental): Japanese participants will be randomized to receive a fixed dose (Dose 1) of vibostolimab in combination with 200 mg pembrolizumab on Day 1 of each 21-day infusion cycle until the 35-cycle limit is reached.
  Interventions: Biological: vibostolimab; Biological: pembrolizumab
- vibostolimab Dose 2 Japanese cohort (Experimental): Japanese participants will be randomized to receive a fixed dose (Dose 2) of vibostolimab in combination with 200 mg pembrolizumab on Day 1 of each 21-day infusion cycle until the 35-cycle limit is reached.
  Interventions: Biological: vibostolimab; Biological: pembrolizumab
- pembrolizumab/vibostolimab coformulation (Experimental): Participants will receive a fixed dose of pembrolizumab/vibostolimab coformulation, consisting of 200 mg of pembrolizumab + 200 mg vibostolimab, on Day 1 of each 21-day infusion cycle for up to 35 cycles.
  Interventions: Biological: pembrolizumab/vibostolimab coformulation
- vibostolimab+pembrolizumab+carboplatin OR cisplatin+etoposide (Experimental): Participants will receive 200 mg vibostolimab in combination with 200 mg pembrolizumab, plus the investigator's choice of Area Under Curve (AUC) 5 mg/mL/min carboplatin OR 75 mg/m^2 cisplatin on Day 1 of each 21-day cycle plus 100 mg/m^2/day etoposide on Days 1-3 of each 21-day cycle for up to 4 cycles. Maintenance therapy with 200 mg vibostolimab in combination with 200 mg pembrolizumab on Day 1 of each 21-day cycle will continue for up to an additional 31 cycles. A participant will be allowed to switch from cisplatin to carboplatin in the event of an adverse event (AE), ineligibility for further cisplatin therapy, and/or the investigator considers switching to carboplatin to be in the best interest of the participant.
  Interventions: Biological: vibostolimab; Biological: pembrolizumab; Drug: carboplatin; Drug: cisplatin; Drug: etoposide
- pembrolizumab/vibostolimab coformulation China cohort (Experimental): Participants from mainland China will receive a fixed dose of pembrolizumab/vibostolimab coformulation, consisting of 200 mg of pembrolizumab + 200 mg vibostolimab, on Day 1 of each 21-day infusion cycle for up to 35 cycles.
  Interventions: Biological: pembrolizumab/vibostolimab coformulation

INTERVENTIONS:
Biological: vibostolimab — Administered as an intravenous (IV) infusion on Day 1 of 21-day infusion Cycles 1-35
  Other Names: MK-7684
  Arms: Advanced solid tumor cohort; Randomized dose 1 comparison cohort; Randomized dose 2 comparison cohort; vibostolimab; vibostolimab + pembrolizumab; vibostolimab +pembrolizumab+pemetrexed+carboplatin; vibostolimab Dose 1 Japanese cohort; vibostolimab Dose 2 Japanese cohort; vibostolimab+pembrolizumab+carboplatin OR cisplatin+etoposide
Biological: pembrolizumab — Administered as an IV infusion on Day 1 of 21-day infusion Cycles 1-35
  Other Names: KEYTRUDA®; MK-3475
  Arms: Advanced solid tumor cohort; Randomized dose 1 comparison cohort; Randomized dose 2 comparison cohort; vibostolimab + pembrolizumab; vibostolimab +pembrolizumab+pemetrexed+carboplatin; vibostolimab Dose 1 Japanese cohort; vibostolimab Dose 2 Japanese cohort; vibostolimab+pembrolizumab+carboplatin OR cisplatin+etoposide
Drug: pemetrexed — Administered as an IV infusion on Day 1 of 21-day infusion Cycles 1-35
  Other Names: ALIMTA®
  Arms: vibostolimab +pembrolizumab+pemetrexed+carboplatin
Drug: carboplatin — Administered as an IV infusion on Day 1 of 21-day infusion Cycles 1-4
  Other Names: PARAPLATIN®
  Arms: vibostolimab +pembrolizumab+pemetrexed+carboplatin; vibostolimab+pembrolizumab+carboplatin OR cisplatin+etoposide
Biological: pembrolizumab/vibostolimab coformulation — Administered as an IV infusion on Day 1 of 21-day infusion Cycles 1-35
  Other Names: MK-7684A
  Arms: pembrolizumab/vibostolimab coformulation; pembrolizumab/vibostolimab coformulation China cohort
Drug: cisplatin — Administered as an IV infusion on Day 1 of 21-day infusion Cycles 1-4
  Other Names: PLATINOL-AQ®
  Arms: vibostolimab+pembrolizumab+carboplatin OR cisplatin+etoposide
Drug: etoposide — Administered as an IV infusion on Days 1-3 of 21-day infusion Cycles 1-4
  Other Names: ETOPOPHOS®
  Arms: vibostolimab+pembrolizumab+carboplatin OR cisplatin+etoposide

SUMMARY:
This is a safety, efficacy, and pharmacokinetics (PK) study of vibostolimab (MK-7684) as monotherapy and in combination with pembrolizumab (MK-3475) or pembrolizumab plus pemetrexed and carboplatin in adults with metastatic solid tumors for which there is no available therapy that is expected to convey clinical benefit. Part A of this study is a dose escalation and confirmation phase to estimate the recommended Phase 2 dose (RPTD) for vibostolimab monotherapy or in combination with pembrolizumab, pemetrexed, and carboplatin. Part A will also evaluate the anti-tumor activity of vibostolimab in combination with pembrolizumab plus pemetrexed and carboplatin in participants with non-small cell lung cancer (NSCLC) and vibostolimab (at two dose levels) in combination with pembrolizumab in Japanese participants with gastric cancer. Part B will evaluate the anti-tumor activity of vibostolimab at the RPTD when used as monotherapy and in combination with pembrolizumab in participants with advanced solid tumors in a non-randomized study design. Part B will also evaluate 2 doses of vibostolimab in combination with pembrolizumab in participants with programmed death 1 (PD-1) treatment naïve cancer using a 1:1 randomized study design. Part B is expanded with Amendment 11 to include an additional arm that will compare the safety and PK of a fixed dose of pembrolizumab/vibostolimab coformulation (MK-7684A) to vibostolimab in combination with pembrolizumab administered as separate intravenous infusions. Part A is expanded with Amendment 12 to include an additional arm that will compare the safety and PK of vibostolimab plus pembrolizumab plus the investigator's choice of platinum agent (carboplatin or cisplatin), and etoposide. Part B is expanded with Amendment 12 to include evaluation of efficacy of vibostolimab plus pembrolizumab plus the investigator's choice of platinum agent (carboplatin or cisplatin), and etoposide and efficacy of pembrolizumab/vibostolimab coformulation in participants from mainland China. The primary hypotheses are that vibostolimab administered as monotherapy or in combination with pembrolizumab is safe and tolerable when administered at the RPTD and that pembrolizumab/vibostolimab coformulation is safe and tolerable when administered as a fixed dose.

ELIGIBILITY:
Inclusion Criteria:

* For Part A participants enrolled prior to Amendment 7, must have a histologically or cytologically confirmed metastatic solid tumor for which there is no available therapy that is expected to convey clinical benefit
* For Part A Japanese cohort added with Amendment 7: Must reside in Japan and be of Japanese descent and have adenocarcinoma of the stomach and/or gastric-esophageal junction (GEJ) that is considered inoperable and that has received, and progressed on, at least 1 prior chemotherapy regimen or human epidermal growth factor receptor 2 (HER2)/neu-targeted approved therapy (if HER2/neu-positive). In both cases, participants may be untreated or could have received and progressed on 1 prior regimen, but must not have received prior anti-PD-1/PD-L1 therapy
* For Part A participants with non-small cell lung cancer (NSCLC) added with Amendment 7: Must have a histologically or cytologically confirmed diagnosis of stage IV (M1a or M1b per current American Joint Committee on Cancer criteria, edition 8) non-squamous NSCLC
* For Part B China participants added with Amendment 12. Must have a histologically or cytologically confirmed metastatic solid tumor for which no more than 2 prior lines of therapy were administered and there is no available therapy that is expected to convey clinical benefit AND be Chinese from mainland China
* For Parts A and B: Has histologically or cytologically confirmed metastatic solid tumor
* Has measurable disease by Response Evaluation Criteria In Solid Tumors (RECIST)
* Has an Eastern Cooperative Oncology Group performance status of 0 to 1
* Females must not be pregnant
* Women of childbearing potential and male participants must agree to use adequate contraception for the course of the study
* Has provided a tumor tissue sample (archival or newly obtained core or excisional biopsy of a tumor lesion)
* For Chinese participants enrolled as part of Amendment 12. No tumor tissue samples will be collected

Exclusion Criteria:

* Has had chemotherapy, radiation, biological cancer therapy or major surgery within 4 weeks prior to the first dose of study treatment
* Has not recovered to Common Toxicity Criteria for Adverse Events Grade 1 or better from the adverse events due to cancer therapeutics administered more than 4 weeks prior to the first dose of study treatment
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment
* Has received previous treatment with another agent targeting the T cell immunoglobulin and immunoreceptor tyrosine-based inhibitory motif (TIGIT) receptor
* Has received previous treatment with an immunomodulatory agent (e.g., anti-programmed cell death 1, anti-programmed cell death ligand 1 or cytotoxic T-lymphocyte-associated protein 4) and was discontinued from that treatment due to a Grade 3 or higher immune-related adverse event
* Is expected to require any other form of antineoplastic therapy while participating in the trial
* Is on chronic systemic steroid therapy in excess of replacement doses or on any other form of immunosuppressive medication
* Has a history of a previous additional malignancy unless potentially curative treatment has been completed with no evidence of malignancy for 5 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has an active autoimmune disease
* Has an active infection requiring systemic treatment
* Has interstitial lung disease
* Has active or past history of (non-infectious) pneumonitis requiring steroids
* Has symptomatic ascites or pleural effusion
* Has previously had a hematopoetic stem cell transplant or solid organ transplant
* Is known to be human immunodeficiency virus (HIV) positive and/or known to have active chronic or acute Hepatitis B or Hepatitis C
* Has a known psychiatric and/or substance abuse disorder that would make it difficult for the participant to cooperate with the requirements of the trial
* Is a regular user (including recreational use) of any illicit drugs at the time of providing documented informed consent, or has a recent history (within the last year) of substance abuse
* Has received a live virus vaccine within 30 days prior to the first dose of study treatment
* Has had hormonal cancer therapy (e.g., tamoxifen, leuprolide). within 4 weeks prior to the first dose of study treatment
* For Part A participants with NSCLC added with Amendment 7: Is unable to interrupt aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs) other than an aspirin dose ≤1.3 gram per day for a 5-day period (8-day period for long-acting agents, such as piroxicam)
* For Part A participants with NSCLC added with Amendment 7: Is unable or unwilling to take folic acid or Vitamin B12 supplementation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Niu J, Maurice-Dror C, Lee DH, Kim DW, Nagrial A, Voskoboynik M, Chung HC, Mileham K, Vaishampayan U, Rasco D, Golan T, Bauer TM, Jimeno A, Chung V, Chartash E, Lala M, Chen Q, Healy JA, Ahn MJ. First-in-human phase 1 study of the anti-TIGIT antibody vibostolimab as monotherapy or with pembrolizumab for advanced solid tumors, including non-small-cell lung cancer☆. Ann Oncol. 2022 Feb;33(2):169-180. doi: 10.1016/j.annonc.2021.11.002. Epub 2021 Nov 18. PMID 34800678
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants at least 18 years of age with advanced solid tumors were enrolled in this study.
Pre-assignment Details: As it was pre-specified to assign treatment groups irrespective of dose level, or cohorts such as based on type of cancer or country of origin, participants were instead combined into treatment groups based on their unique combination of interventions. For dose escalation, it was pre-specifed that participants were combined into monotherapy or sequential treatment groups rather than separate dose levels. Parts A and B were conducted at the same time, not sequentially.
Groups:
- Vibostolimab: During an initial dose evaluation phase, participants received various doses of vibostolimab on Day 1 of each 21-day infusion cycle (for a maximum of 35 cycles) until the recommended Phase 2 dose (RPTD) of 200 mg was established based on the number of dose limiting toxicities (DLTs) at each dose level. Participants continued receiving 200 mg vibostolimab on Day 1 of each 21-day infusion cycle until the 35-cycle limit is reached.
- Vibostolimab + Pembrolizumab: During an initial dose evaluation phase, participants received various doses of vibostolimab in combination with 200 mg pembrolizumab on Day 1 of each 21-day infusion cycle (for a maximum of 35 cycles) until the RPTD of vibostolimab of 200 mg was established based on the number of DLTs at each dose level. Participants continued receiving 200 mg of vibostolimab in combination with 200 mg pembrolizumab on Day 1 of each 21-day infusion cycle until the 35-cycle limit was reached.
- Pembrolizumab/Vibostolimab Coformulation (MK-7684A): Participants received a fixed dose of pembrolizumab/vibostolimab coformulation, consisting of 200 mg of pembrolizumab + 200 mg vibostolimab, on Day 1 of each 21-day infusion cycle for up to 35 cycles.
- Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin: Participants received a 200 mg dose of vibostolimab in combination with 200 mg pembrolizumab, 500 mg/m^2 pemetrexed, and Area Under Curve (AUC) 5 mg/mL/min carboplatin on Day 1 of each 21-day infusion cycle for up to 4 cycles followed by maintenance therapy with a 200 mg dose of vibostolimab in combination with 200 mg pembrolizumab and 500 mg/m^2 pemetrexed on Day 1 of each 21-day infusion cycle for up to an additional 31 cycles.
- Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide: Participants received 200 mg vibostolimab in combination with 200 mg pembrolizumab, plus the investigator's choice of Area Under Curve (AUC) 5 mg/mL/min carboplatin OR 75 mg/m^2 cisplatin on Day 1 of each 21-day cycle plus 100 mg/m^2/day etoposide on Days 1-3 of each 21-day cycle for up to 4 cycles. Maintenance therapy with 200 mg vibostolimab in combination with 200 mg pembrolizumab on Day 1 of each 21-day cycle will continue for up to an additional 31 cycles. A participant will be allowed to switch from cisplatin to carboplatin in the event of an adverse event (AE), ineligibility for further cisplatin therapy, and/or the investigator considers switching to carboplatin to be in the best interest of the participant.
Period: Overall Study
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide
Started (Randomized) | 68 | 295 | 60 | 11 | 40
Treated | 68 | 293 | 60 | 10 | 40
Crossed Over | 25 (Crossed over from vibostolimab monotherapy to vibostolimab + pembrolizumab as sequential administration.) | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 68 | 295 | 60 | 11 | 40
Not completed — Death | 58 | 239 | 38 | 10 | 33
Not completed — Lost to Follow-up | 1 | 4 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0
Not completed — Sponsor Decision | 3 | 22 | 11 | 0 | 7
Not completed — Withdrawal by Subject | 6 | 27 | 9 | 0 | 0
Not completed — Not Treated | 0 | 2 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The population analyzed was treated participants. As it was pre-specified to assign treatment groups irrespective of dose level, or cohorts such as based on type of cancer or country of origin, participants were instead combined into treatment groups based on their unique combination of interventions. For dose escalation, it was pre-specifed that participants were combined into monotherapy or sequential treatment groups rather than separate dose levels
Groups:
- Total: Total of all reporting groups
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide | Total
Number analyzed (Participants) | 68 | 293 | 60 | 10 | 40 | 471
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.1 (12.0) | 57.6 (12.0) | 58.5 (10.0) | 68.5 (9.0) | 66.2 (8.2) | 59.3 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 190 | 43 | 5 | 10 | 282
  Male | 34 | 103 | 17 | 5 | 30 | 189
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 17 | 1 | 0 | 2 | 27
  Not Hispanic or Latino | 59 | 268 | 57 | 9 | 37 | 430
  Unknown or Not Reported | 2 | 8 | 2 | 1 | 1 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 13 | 99 | 25 | 5 | 27 | 169
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 8 | 1 | 0 | 0 | 16
  White | 48 | 181 | 34 | 5 | 12 | 280
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 5 | 0 | 0 | 1 | 6

OUTCOME MEASURES:

1. Secondary Outcome: Overall Response Rate (ORR) in Participants in Vibostolimab Dose Escalation Phase Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: ORR is the percentage of participants who experience complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions) at any time during the trial using RECIST, version 1.1 as assessed by investigator review. Results for participants treated with vibostolimab dose escalation are presented.
Time Frame: Up to 24 Months
Population: Participants with a baseline scan with measurable disease by investigator assessment who were administered a dose of study treatment regardless of dose level. Only dose escalation treatment groups were analyzed, who were assigned based on their combination of interventions rather than by dosage levels.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Vibostolimab + Pembrolizumab After Crossover: After discontinuing vibostolimab monotherapy due to progressive disease participants who crossed over to vibostolimab + pembrolizumab as sequential administration.
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Vibostolimab + Pembrolizumab After Crossover | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide
Number analyzed (Participants) | 34 | 42 | 0 | 0 | 0 | 0
Percentage of participants | 0.0 [0.0 to 10.3] | 7.1 [1.5 to 19.5] |  |  |  |

2. Secondary Outcome: ORR in Participants With Programmed Death 1 (PD-1) Refractory Non-small Cell Lung Cancer (NSCLC) Per RECIST 1.1
Description: ORR is the percentage of participants who experience complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions) at any time during the trial using RECIST, version 1.1 as assessed by investigator review. Results for participants with PD-1 refractory NSCLC treated with 200 or 210 mg vibostolimab in dose escalation as well as dose expansion phases are presented.
Time Frame: Up to 24 Months
Population: Participants with a baseline scan with measurable disease by investigator assessment who were administered a dose of study treatment regardless of dose level. Both dose escalation and expansion phases were analyzed, assigned to treatment groups based on their combination of interventions rather than by dosage levels.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Vibostolimab + Pembrolizumab After Crossover | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide
Number analyzed (Participants) | 41 | 38 | 0 | 0 | 0 | 0
Percentage of participants | 2.4 [0.1 to 12.9] | 5.3 [0.6 to 17.7] |  |  |  |

3. Secondary Outcome: ORR in Participants With PD-1 Naive NSCLC Per RECIST 1.1
Description: ORR is the percentage of participants who experience complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions) at any time during the trial using RECIST, version 1.1 as assessed by investigator review. Results for participants with PD-1 naive NSCLC treated with pembrolizumab and 200 mg vibostolimab from both the dose escalation and expansion phases are presented.
Time Frame: Up to 24 Months
Population: Participants with a baseline scan with measurable disease by investigator assessment who were administered a dose of study treatment regardless of dose level. Both dose escalation and expansion phases were analyzed assigned to treatment groups based on their combination of interventions rather than by dosage levels.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Vibostolimab + Pembrolizumab After Crossover | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide
Number analyzed (Participants) | 0 | 41 | 0 | 0 | 0 | 0
Percentage of participants |  | 24.4 [12.4 to 40.3] |  |  |  |

4. Secondary Outcome: ORR in Participants With Extensive-stage Small Cell Lung Cancer (ES-SCLC) Per RECIST 1.1
Description: ORR is the percentage of participants who experience complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions) at any time during the trial using RECIST, version 1.1 as assessed by investigator review. Participants with ES-SCLC treated with vibostolimab in combination with pembrolizumab, carboplatin or cisplatin, and etoposide were analyzed.
Time Frame: Up to 24 Months
Population: Participants with a baseline scan with measurable disease by investigator assessment who were administered a dose of study treatment regardless of dose level. For ES-SCLC only participants in the etoposide treatment group were analyzed, based on their combination of interventions rather than by dosage levels.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Vibostolimab + Pembrolizumab After Crossover | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 40
Percentage of participants |  |  |  |  |  | 75.0 [58.8 to 87.3]

5. Secondary Outcome: ORR in Participants With PD-1 Naive Ovarian Cancer Per RECIST 1.1
Description: ORR is the percentage of participants who experience complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions) at any time during the trial using RECIST, version 1.1 as assessed by investigator review. Participants with PD-1 naive ovarian cancer treated with pembrolizumab and vibostolimab dose escalation or MK-7984A were analyzed.
Time Frame: Up to 24 Months
Population: Participants with a baseline scan with measurable disease by investigator assessment who were administered a dose of study treatment regardless of dose level. For PD-1 naive ovarian cancer only participants treated with vibostolimab and pembrolizumab taken sequentially, or as a coformulation were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Vibostolimab + Pembrolizumab After Crossover | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide
Number analyzed (Participants) | 0 | 21 | 0 | 40 | 0 | 0
Percentage of participants |  | 9.5 [1.2 to 30.4] |  | 7.5 [1.6 to 20.4] |  |

6. Secondary Outcome: ORR in Participants With PD-1 Naive Cervical Cancer Per RECIST 1.1
Description: ORR is the percentage of participants who experience complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions) at any time during the trial using RECIST, version 1.1 as assessed by investigator review. Results for participants with PD-1 naive cervical cancer treated with pembrolizumab and either 200 mg or 700 mg vibostolimab are presented.
Time Frame: Up to 24 Months
Population: Participants with a baseline scan with measurable disease by investigator assessment who were administered a dose of study treatment regardless of dose level. For PD-1 naive cervical cancer only participants treated with vibostolimab and pembrolizumab sequentially were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Vibostolimab + Pembrolizumab After Crossover | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide
Number analyzed (Participants) | 0 | 41 | 0 | 0 | 0 | 0
Percentage of participants
  Vibostolimab 200 mg |  | 14.6 [5.6 to 29.2] |  |  |  |
  Vibostolimab 700 mg: number analyzed (Participants) | 0 | 39 | 0 | 0 | 0 | 0
  Vibostolimab 700 mg |  | 23.1 [11.1 to 39.3] |  |  |  |

7. Secondary Outcome: Area Under the Curve From Time 0 to 21 Days Postdose (AUC 0-21 Days) of Plasma Vibostolimab Following Treatment With Increasing Amounts of Vibostolimab Monotherapy or Vibostolimab With 200 mg Pembrolizumab
Description: Blood samples were collected from participants during cycle 1 and cycle 4 of treatment (Cycle length is 21 days) in order to determine the AUC 0-21 days of plasma vibostolimab, Only results from participants treated with increasing amounts of vibostolimab monotherapy or vibostolimab combined with 200 mg pembrolizumab are presented; whereas other treatment groups were not analyzed. Due to terminal fitting issue, non-calculable AUC0-21 days was replaced with AUClast for a few participants.
Time Frame: Cycle 1, Cycle 4: Day 1 pre-dose, 0.5, and 2 hours post-dose; once daily on Days 2, 3, 5, 8, 15 and 22.
Population: Participants who complied with the protocol sufficiently to ensure that the data they generated will be likely to exhibit the effects of treatment, according to the underlying scientific model. Compliance covers such considerations as exposure to treatment, availability of measurements, and absence of major protocol violations. Only participants with dose escalation were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: day*μg/mL
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Vibostolimab + Pembrolizumab After Crossover | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide
Number analyzed (Participants) | 48 | 230 | 0 | 0 | 0 | 0
day*μg/mL
  Vibostolimab 2.10 mg Cycle 1: number analyzed (Participants) | 3 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 2.10 mg Cycle 1 | 5.42 [0.209 to 141] | 8.19 [0.267 to 252] |  |  |  |
  Vibostolimab 7.00 mg Cycle 1: number analyzed (Participants) | 3 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 7.00 mg Cycle 1 | 12.2 [6.58 to 22.7] | 12.0 [0.0276 to 5240] |  |  |  |
  Vibostolimab 7.00 mg Cycle 4: number analyzed (Participants) | 3 | 1 | 0 | 0 | 0 | 0
  Vibostolimab 7.00 mg Cycle 4 | 12.4 [3.75 to 41.0] | NA [NA to NA] — Due to insufficient data, results were not analyzed |  |  |  |
  Vibostolimab 21.0 mg Cycle 1: number analyzed (Participants) | 3 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 21.0 mg Cycle 1 | 38.3 [23.2 to 63.3] | 28.5 [7.54 to 107] |  |  |  |
  Vibostolimab 21.0 mg Cycle 4: number analyzed (Participants) | 1 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 21.0 mg Cycle 4 | NA [NA to NA] — Due to insufficient data, results were not analyzed | 48.3 [30.9 to 75.5] |  |  |  |
  Vibostolimab 70.0 mg Cycle 1: number analyzed (Participants) | 4 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 70.0 mg Cycle 1 | 97.7 [24.4 to 391] | 156 [78.6 to 308] |  |  |  |
  Vibostolimab 200 mg Cycle 1 | 339 [306 to 377] | 354 [338 to 371] |  |  |  |
  Vibostolimab 200 mg Cycle 4: number analyzed (Participants) | 18 | 124 | 0 | 0 | 0 | 0
  Vibostolimab 200 mg Cycle 4 | 572 [478 to 685] | 519 [475 to 568] |  |  |  |
  Vibostolimab 700 mg Cycle 1: number analyzed (Participants) | 7 | 49 | 0 | 0 | 0 | 0
  Vibostolimab 700 mg Cycle 1 | 1220 [828 to 1800] | 1250 [1120 to 1400] |  |  |  |
  Vibostolimab 700 mg Cycle 4: number analyzed (Participants) | 4 | 26 | 0 | 0 | 0 | 0
  Vibostolimab 700 mg Cycle 4 | 1090 [273 to 4380] | 2080 [1800 to 2410] |  |  |  |

8. Secondary Outcome: AUC 0-21 Days of Plasma Vibostolimab Following Treatment With 200 mg Vibostolimab Combined With Various Other Treatments
Description: Blood samples were collected from participants during cycle 1 and cycle 4 of treatment (Cycle length is 21 days) following treatment with 200 mg vibostolimab in order to determine the AUC 0-21 days of plasma vibostolimab, Due to terminal fitting issue, non-calculable AUC0-21 days was replaced with AUClast for a few participants.
Time Frame: Cycle 1, Cycle 4: Day 1 pre-dose, 0.5 and 2 hours post-dose; once daily on Days 2, 3, 5, 8, 15 and 22
Population: Participants who complied with the protocol sufficiently to ensure that the data they generated will be likely to exhibit the effects of treatment, according to the underlying scientific model. Compliance covers such considerations as exposure to treatment, availability of measurements, and absence of major protocol violations. Cycle 4 for participants treated with etoposide was not analyzed due to insufficient time points available to determine AUC0-21 days.
Measure: Geometric Mean (95% Confidence Interval); unit: day*μg/mL
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Vibostolimab + Pembrolizumab After Crossover | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide
Number analyzed (Participants) | 48 | 230 | 0 | 60 | 10 | 38
day*μg/mL
  200 mg vibostolimab Cycle 1 | 339 [306 to 377] | 354 [338 to 371] |  | 431 [398 to 466] | 317 [267 to 378] | 476 [417 to 543]
  200 mg vibostolimab Cycle 4: number analyzed (Participants) | 18 | 124 | 0 | 19 | 8 | 0
  200 mg vibostolimab Cycle 4 | 572 [478 to 685] | 519 [475 to 568] |  | 655 [510 to 843] | 342 [166 to 703] |

9. Secondary Outcome: AUC 0-21 Days of Plasma Pembrolizumab Following Treatment With Increasing Amounts of Vibostolimab With 200 mg Pembrolizumab
Description: Blood samples were collected from participants during cycle 1 and cycle 4 of treatment (Cycle length is 21 days) in order to determine the AUC 0-21 days of plasma vibostolimab, Only results from participants treated with increasing amounts of vibostolimab combined with 200 mg pembrolizumab are presented; whereas other treatment groups were not analyzed. Due to terminal fitting issue, non-calculable AUC0-21 days was replaced with AUClast for a few participants.
Time Frame: Cycle 1, Cycle 4: Day 1 pre-dose, 0.5 and 2 hours post-dose; once daily on Days 2, 3, 5, 8, 15 and 22
Population: Participants who complied with the protocol sufficiently to ensure that the data they generated will be likely to exhibit the effects of treatment, according to the underlying scientific model. Compliance covers such considerations as exposure to treatment, availability of measurements, and absence of major protocol violations. Only participants with pembrolizumab and dose escalation were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: day*μg/mL
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Vibostolimab + Pembrolizumab After Crossover | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide
Number analyzed (Participants) | 0 | 229 | 0 | 0 | 0 | 0
day*μg/mL
  Vibostolimab 2.10 mg Cycle 1: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 2.10 mg Cycle 1 |  | 760 [650 to 888] |  |  |  |
  Vibostolimab 7.00 mg Cycle 1: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 7.00 mg Cycle 1 |  | 749 [457 to 1230] |  |  |  |
  Vibostolimab 7.00 mg Cycle 4: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Vibostolimab 7.00 mg Cycle 4 |  | NA [NA to NA] — Due to insufficient data, results were not analyzed |  |  |  |
  Vibostolimab 21.0 mg Cycle 1: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 21.0 mg Cycle 1 |  | 516 [211 to 1260] |  |  |  |
  Vibostolimab 21.0 mg Cycle 4: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 21.0 mg Cycle 4 |  | 922 [626 to 1360] |  |  |  |
  Vibostolimab 70.0 mg Cycle 1: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 70.0 mg Cycle 1 |  | 504 [321 to 792] |  |  |  |
  Vibostolimab 200 mg Cycle 1 |  | 516 [497 to 535] |  |  |  |
  Vibostolimab 200 mg Cycle 4: number analyzed (Participants) | 0 | 124 | 0 | 0 | 0 | 0
  Vibostolimab 200 mg Cycle 4 |  | 887 [838 to 938] |  |  |  |
  Vibostolimab 700 mg Cycle 1: number analyzed (Participants) | 0 | 49 | 0 | 0 | 0 | 0
  Vibostolimab 700 mg Cycle 1 |  | 541 [496 to 589] |  |  |  |
  Vibostolimab 700 mg Cycle 4: number analyzed (Participants) | 0 | 26 | 0 | 0 | 0 | 0
  Vibostolimab 700 mg Cycle 4 |  | 1050 [912 to 1210] |  |  |  |

10. Secondary Outcome: AUC 0-21 Days of Plasma Pembrolizumab Following Treatment With 200 mg Vibostolimab and 200 mg Pembrolizumab Combined With Various Other Treatments
Description: Blood samples were collected from participants during cycle 1 and cycle 4 of treatment (Cycle length is 21 days) following treatment with 200 mg vibostolimab and 200 mg pembrolizumab in order to determine the AUC 0-21 days of plasma pembrolizumab. Due to terminal fitting issue, non-calculable AUC0-21 days was replaced with AUClast for a few participants.
Time Frame: Cycle 1, Cycle 4: Day 1 pre-dose, 0.5 and 2 hours post-dose; once daily on Days 2, 3, 5, 8, 15 and 22
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: day*μg/mL
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Vibostolimab + Pembrolizumab After Crossover | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide
Number analyzed (Participants) | 0 | 229 | 0 | 60 | 10 | 39
day*μg/mL
  Cycle 1 |  | 516 [497 to 535] |  | 546 [507 to 588] | 539 [473 to 615] | 641 [601 to 682]
  Cycle 4: number analyzed (Participants) | 0 | 124 | 0 | 19 | 8 | 0
  Cycle 4 |  | 887 [838 to 938] |  | 946 [765 to 1170] | 974 [815 to 1160] |

11. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Plasma Vibostolimab Following Treatment With Increasing Amounts of Vibostolimab Monotherapy or Vibostolimab With 200 mg Pembrolizumab
Description: Blood samples were collected from participants during cycle 1 and cycle 4 of treatment (Cycle length is 21 days) in order to determine the Cmax of plasma vibostolimab, Only results from participants treated with increasing amounts of vibostolimab monotherapy or vibostolimab combined with 200 mg pembrolizumab are presented; whereas other treatment groups were not analyzed.
Time Frame: Cycle 1, Cycle 4: Day 1 pre-dose, 0.5 and 2 hours post-dose; once daily on Days 2, 3, 5, 8, 15 and 22
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Vibostolimab + Pembrolizumab After Crossover | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide
Number analyzed (Participants) | 48 | 230 | 0 | 0 | 0 | 0
μg/mL
  Vibostolimab 2.10 mg Cycle 1: number analyzed (Participants) | 3 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 2.10 mg Cycle 1 | 1.52 [0.173 to 13.4] | 1.67 [0.114 to 24.5] |  |  |  |
  Vibostolimab 7.00 mg Cycle 1: number analyzed (Participants) | 3 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 7.00 mg Cycle 1 | 7.23 [0.914 to 57.2] | 2.09 [1.01 to 4.34] |  |  |  |
  Vibostolimab 7.00 mg Cycle 4: number analyzed (Participants) | 3 | 1 | 0 | 0 | 0 | 0
  Vibostolimab 7.00 mg Cycle 4 | 7.57 [0.266 to 215] | NA [NA to NA] — Due to insufficient data, results were not analyzed |  |  |  |
  Vibostolimab 21.0 mg Cycle 1: number analyzed (Participants) | 3 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 21.0 mg Cycle 1 | 8.64 [6.73 to 11.1] | 4.70 [1.48 to 14.9] |  |  |  |
  Vibostolimab 21.0 mg Cycle 4: number analyzed (Participants) | 1 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 21.0 mg Cycle 4 | NA [NA to NA] — Due to insufficient data, results were not analyzed | 6.30 [4.22 to 9.40] |  |  |  |
  Vibostolimab 70.0 mg Cycle 1: number analyzed (Participants) | 4 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 70.0 mg Cycle 1 | 19.5 [11.8 to 32.3] | 24.9 [18.5 to 33.5] |  |  |  |
  Vibostolimab 200 mg Cycle 1 | 62.6 [56.4 to 69.4] | 64.4 [60.8 to 68.2] |  |  |  |
  Vibostolimab 200 mg Cycle 4: number analyzed (Participants) | 18 | 124 | 0 | 0 | 0 | 0
  Vibostolimab 200 mg Cycle 4 | 82.7 [70.0 to 97.8] | 80.1 [72.9 to 87.9] |  |  |  |
  Vibostolimab 700 mg Cycle 1: number analyzed (Participants) | 7 | 49 | 0 | 0 | 0 | 0
  Vibostolimab 700 mg Cycle 1 | 202 [165 to 248] | 236 [209 to 266] |  |  |  |
  Vibostolimab 700 mg Cycle 4: number analyzed (Participants) | 4 | 26 | 0 | 0 | 0 | 0
  Vibostolimab 700 mg Cycle 4 | 215 [137 to 337] | 245 [217 to 276] |  |  |  |

12. Secondary Outcome: Cmax of Plasma Vibostolimab Following Treatment With 200 mg Vibostolimab Combined With Various Other Treatments
Description: Blood samples were collected from participants during cycle 1 and cycle 4 of treatment (Cycle length is 21 days) following treatment with 200 mg vibostolimab in order to determine the Cmax of plasma vibostolimab,
Time Frame: Cycle 1, Cycle 4: Day 1 pre-dose, 0.5 and 2 hours post-dose; once daily on Days 2, 3, 5, 8, 15 and 22
Population: Participants who complied with the protocol sufficiently to ensure that the data they generated will be likely to exhibit the effects of treatment, according to the underlying scientific model. Compliance covers such considerations as exposure to treatment, availability of measurements, and absence of major protocol violations. Cycle 4 for participants treated with etoposide was not analyzed due to insufficient time points available to determine Cmax.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Vibostolimab + Pembrolizumab After Crossover | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide
Number analyzed (Participants) | 48 | 230 | 0 | 60 | 10 | 38
μg/mL
  200 mg vibostolimab Cycle 1 | 62.6 [56.4 to 69.4] | 64.4 [60.8 to 68.2] |  | 59.9 [55.0 to 65.2] | 60.1 [51.6 to 70.1] | 59.6 [51.9 to 68.4]
  200 mg vibostolimab Cycle 4: number analyzed (Participants) | 18 | 124 | 0 | 19 | 8 | 0
  200 mg vibostolimab Cycle 4 | 82.7 [70.0 to 97.8] | 80.1 [72.9 to 87.9] |  | 56.4 [44.2 to 72.0] | 57.8 [45.5 to 73.5] |

13. Secondary Outcome: Cmax of Plasma Pembrolizumab Following Treatment With Increasing Amounts of Vibostolimab With 200 mg Pembrolizumab
Description: Blood samples were collected from participants during cycle 1 and cycle 4 of treatment (Cycle length is 21 days) in order to determine the Cmax of plasma vibostolimab, Only results from participants treated with increasing amounts of vibostolimab combined with 200 mg pembrolizumab are presented; whereas other treatment groups were not analyzed.
Time Frame: Cycle 1, Cycle 4: Day 1 pre-dose, 0.5 and 2 hours post-dose; once daily on Days 2, 3, 5, 8, 15 and 22
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Vibostolimab + Pembrolizumab After Crossover | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide
Number analyzed (Participants) | 0 | 229 | 0 | 0 | 0 | 0
μg/mL
  Vibostolimab 2.10 mg Cycle 1: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 2.10 mg Cycle 1 |  | 89.3 [76.6 to 104] |  |  |  |
  Vibostolimab 7.00 mg Cycle 1: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 7.00 mg Cycle 1 |  | 86.4 [35.9 to 208] |  |  |  |
  Vibostolimab 7.00 mg Cycle 4: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Vibostolimab 7.00 mg Cycle 4 |  | NA [NA to NA] — Due to insufficient data, results were not analyzed |  |  |  |
  Vibostolimab 21.0 mg Cycle 1: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 21.0 mg Cycle 1 |  | 58.4 [29.3 to 116] |  |  |  |
  Vibostolimab 21.0 mg Cycle 4: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 21.0 mg Cycle 4 |  | 95.0 [84.4 to 107] |  |  |  |
  Vibostolimab 70.0 mg Cycle 1: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 70.0 mg Cycle 1 |  | 90.5 [79.9 to 103] |  |  |  |
  Vibostolimab 200 mg Cycle 1 |  | 76.1 [73.7 to 78.6] |  |  |  |
  Vibostolimab 200 mg Cycle 4: number analyzed (Participants) | 0 | 124 | 0 | 0 | 0 | 0
  Vibostolimab 200 mg Cycle 4 |  | 93.9 [89.3 to 98.6] |  |  |  |
  Vibostolimab 700 mg Cycle 1: number analyzed (Participants) | 0 | 49 | 0 | 0 | 0 | 0
  Vibostolimab 700 mg Cycle 1 |  | 81.6 [74.6 to 89.3] |  |  |  |
  Vibostolimab 700 mg Cycle 4: number analyzed (Participants) | 0 | 26 | 0 | 0 | 0 | 0
  Vibostolimab 700 mg Cycle 4 |  | 103 [94.7 to 113] |  |  |  |

14. Secondary Outcome: Cmax of Plasma Pembrolizumab Following Treatment With 200 mg Vibostolimab and 200 mg Pembrolizumab Combined With Various Other Treatments
Description: Blood samples were collected from participants during cycle 1 and cycle 4 of treatment (Cycle length is 21 days) following treatment with 200 mg vibostolimab and 200 mg pembrolizumab in order to determine the Cmax of plasma pembrolizumab.
Time Frame: Cycle 1, Cycle 4: Day 1 pre-dose, 0.5 and 2 hours post-dose; once daily on Days 2, 3, 5, 8, 15 and 22
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Vibostolimab + Pembrolizumab After Crossover | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide
Number analyzed (Participants) | 0 | 229 | 0 | 60 | 10 | 39
μg/mL
  Cycle 1 |  | 76.1 [73.7 to 78.6] |  | 66.4 [60.6 to 72.8] | 71.6 [63.2 to 81.2] | 64.4 [60.6 to 68.4]
  Cycle 4: number analyzed (Participants) | 0 | 124 | 0 | 19 | 8 | 0
  Cycle 4 |  | 93.9 [89.3 to 98.6] |  | 73.2 [60.4 to 88.6] | 91.1 [78.6 to 106] |

15. Secondary Outcome: Trough Concentration (Ctrough) of Plasma Vibostolimab Following Treatment With Increasing Amounts of Vibostolimab Monotherapy or Vibostolimab With 200 mg Pembrolizumab
Description: Blood samples were collected from participants during cycle 1 and cycle 4 of treatment (Cycle length is 21 days) in order to determine the Ctrough of plasma vibostolimab, Only results from participants treated with increasing amounts of vibostolimab monotherapy or vibostolimab combined with 200 mg pembrolizumab are presented; whereas other treatment groups were not analyzed.
Time Frame: Cycle 1, Cycle 4: Day 1 pre-dose, 0.5 and 2 hours post-dose; once daily on Days 2, 3, 5, 8, 15 and 22
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Vibostolimab + Pembrolizumab After Crossover | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide
Number analyzed (Participants) | 48 | 230 | 0 | 0 | 0 | 0
μg/mL
  Vibostolimab 2.10 mg Cycle 1: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0
  Vibostolimab 2.10 mg Cycle 1 | NA [NA to NA] — Insufficient timepoints available to determine Ctrough | NA [NA to NA] — Insufficient timepoints available to determine Ctrough |  |  |  |
  Vibostolimab 7.00 mg Cycle 1: number analyzed (Participants) | 3 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 7.00 mg Cycle 1 | NA [NA to NA] — Insufficient timepoints available to calculate | NA [NA to NA] — Insufficient timepoints available to calculate |  |  |  |
  Vibostolimab 7.00 mg Cycle 4: number analyzed (Participants) | 3 | 1 | 0 | 0 | 0 | 0
  Vibostolimab 7.00 mg Cycle 4 | NA [NA to NA] — Insufficient timepoints available to calculate | NA [NA to NA] — Insufficient timepoints available to determine Ctrough |  |  |  |
  Vibostolimab 21.0 mg Cycle 1: number analyzed (Participants) | 3 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 21.0 mg Cycle 1 | 0.539 [0.213 to 1.36] | 0.397 [0.0719 to 2.19] |  |  |  |
  Vibostolimab 21.0 mg Cycle 4: number analyzed (Participants) | 1 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 21.0 mg Cycle 4 | NA [NA to NA] — Insufficient timepoints available to determine Ctrough | 1.11 [0.698 to 1.76] |  |  |  |
  Vibostolimab 70.0 mg Cycle 1: number analyzed (Participants) | 4 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 70.0 mg Cycle 1 | 3.21 [0.623 to 16.5] | 1.79 [0.240 to 13.3] |  |  |  |
  Vibostolimab 200 mg Cycle 1 | 3.82 [2.62 to 5.57] | 5.05 [4.43 to 5.76] |  |  |  |
  Vibostolimab 200 mg Cycle 4: number analyzed (Participants) | 18 | 124 | 0 | 0 | 0 | 0
  Vibostolimab 200 mg Cycle 4 | 10.7 [6.73 to 17.1] | 9.66 [8.03 to 11.6] |  |  |  |
  Vibostolimab 700 mg Cycle 1: number analyzed (Participants) | 7 | 49 | 0 | 0 | 0 | 0
  Vibostolimab 700 mg Cycle 1 | 10.0 [0.929 to 108] | 19.3 [15.2 to 24.6] |  |  |  |
  Vibostolimab 700 mg Cycle 4: number analyzed (Participants) | 4 | 26 | 0 | 0 | 0 | 0
  Vibostolimab 700 mg Cycle 4 | 41.3 [10.1 to 169] | 40.1 [28.2 to 57.0] |  |  |  |

16. Secondary Outcome: Ctrough of Plasma Vibostolimab Following Treatment With 200 mg Vibostolimab Combined With Various Other Treatments
Description: Blood samples were collected from participants during cycle 1 and cycle 4 of treatment (Cycle length is 21 days) following treatment with 200 mg vibostolimab in order to determine the Ctrough of plasma vibostolimab,
Time Frame: Cycle 1, Cycle 4: Day 1 pre-dose, 0.5 and 2 hours post-dose; once daily on Days 2, 3, 5, 8, 15 and 22
Population: Participants who complied with the protocol sufficiently to ensure that the data they generated will be likely to exhibit the effects of treatment, according to the underlying scientific model. Compliance covers such considerations as exposure to treatment, availability of measurements, and absence of major protocol violations. Cycle 4 for participants treated with etoposide was not analyzed due to insufficient time points available to determine Ctrough.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Vibostolimab + Pembrolizumab After Crossover | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide
Number analyzed (Participants) | 48 | 230 | 0 | 60 | 10 | 38
μg/mL
  200 mg vibostolimab Cycle 1 | 3.82 [2.62 to 5.57] | 5.05 [4.43 to 5.76] |  | 8.01 [7.16 to 8.97] | 2.50 [1.10 to 5.69] | 4.16 [3.16 to 5.48]
  200 mg vibostolimab Cycle 4: number analyzed (Participants) | 18 | 124 | 0 | 19 | 8 | 0
  200 mg vibostolimab Cycle 4 | 10.7 [6.73 to 17.1] | 9.66 [8.03 to 11.6] |  | 15.5 [11.7 to 20.6] | 9.01 [4.24 to 19.1] |

17. Secondary Outcome: Ctrough of Plasma Pembrolizumab Following Treatment With Increasing Amounts of Vibostolimab With 200 mg Pembrolizumab
Description: Blood samples were collected from participants during cycle 1 and cycle 4 of treatment (Cycle length is 21 days) in order to determine the Ctrough of plasma vibostolimab, Only results from participants treated with increasing amounts of vibostolimab combined with 200 mg pembrolizumab are presented; whereas other treatment groups were not analyzed.
Time Frame: Cycle 1, Cycle 4: Day 1 pre-dose, 0.5 and 2 hours post-dose; once daily on Days 2, 3, 5, 8, 15 and 22
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Vibostolimab + Pembrolizumab After Crossover | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide
Number analyzed (Participants) | 0 | 229 | 0 | 0 | 0 | 0
μg/mL
  Vibostolimab 2.10 mg Cycle 1: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 2.10 mg Cycle 1 |  | 19.8 [17.5 to 22.4] |  |  |  |
  Vibostolimab 7.00 mg Cycle 1: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 7.00 mg Cycle 1 |  | 20.6 [12.4 to 34.1] |  |  |  |
  Vibostolimab 7.00 mg Cycle 4: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Vibostolimab 7.00 mg Cycle 4 |  | NA [NA to NA] — Due to insufficient data, results were not analyzed |  |  |  |
  Vibostolimab 21.0 mg Cycle 1: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 21.0 mg Cycle 1 |  | 10.4 [3.27 to 33.0] |  |  |  |
  Vibostolimab 21.0 mg Cycle 4: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 21.0 mg Cycle 4 |  | 28.0 [17.6 to 44.5] |  |  |  |
  Vibostolimab 70.0 mg Cycle 1: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 70.0 mg Cycle 1 |  | 12.3 [7.10 to 21.4] |  |  |  |
  Vibostolimab 200 mg Cycle 1 |  | 12.1 [11.4 to 12.9] |  |  |  |
  Vibostolimab 200 mg Cycle 4: number analyzed (Participants) | 0 | 124 | 0 | 0 | 0 | 0
  Vibostolimab 200 mg Cycle 4 |  | 23.3 [21.4 to 25.3] |  |  |  |
  Vibostolimab 700 mg Cycle 1: number analyzed (Participants) | 0 | 49 | 0 | 0 | 0 | 0
  Vibostolimab 700 mg Cycle 1 |  | 11.1 [9.31 to 13.3] |  |  |  |
  Vibostolimab 700 mg Cycle 4: number analyzed (Participants) | 0 | 26 | 0 | 0 | 0 | 0
  Vibostolimab 700 mg Cycle 4 |  | 25.7 [18.9 to 35.1] |  |  |  |

18. Secondary Outcome: Ctrough of Plasma Pembrolizumab Following Treatment With 200 mg Vibostolimab and 200 mg Pembrolizumab Combined With Various Other Treatments
Description: Blood samples were collected from participants during cycle 1 and cycle 4 of treatment (Cycle length is 21 days) following treatment with 200 mg vibostolimab and 200 mg pembrolizumab in order to determine the Ctrough of plasma pembrolizumab.
Time Frame: Cycle 1, Cycle 4: Day 1 pre-dose, 0.5 and 2 hours post-dose; once daily on Days 2, 3, 5, 8, 15 and 22
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Vibostolimab + Pembrolizumab After Crossover | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide
Number analyzed (Participants) | 0 | 229 | 0 | 60 | 10 | 39
μg/mL
  Cycle 1 |  | 12.1 [11.4 to 12.9] |  | 13.2 [12.1 to 14.3] | 12.5 [8.98 to 17.3] | 10.9 [10.1 to 11.8]
  Cycle 4: number analyzed (Participants) | 0 | 124 | 0 | 19 | 8 | 0
  Cycle 4 |  | 23.3 [21.4 to 25.3] |  | 24.7 [19.4 to 31.3] | 31.0 [23.3 to 41.1] |

19. Secondary Outcome: Half Life (t1/2)) of Plasma Vibostolimab Following Treatment With Increasing Amounts of Vibostolimab Monotherapy or Vibostolimab With 200 mg Pembrolizumab
Description: Blood samples were collected from participants during cycle 1 and cycle 4 of treatment (Cycle length is 21 days) in order to determine the t1/2 of plasma vibostolimab, Only results from participants treated with increasing amounts of vibostolimab monotherapy or vibostolimab combined with 200 mg pembrolizumab are presented; whereas other treatment groups were not analyzed.
Time Frame: Cycle 1, Cycle 4: Day 1 pre-dose, 0.5 and 2 hours post-dose; once daily on Days 2, 3, 5, 8, 15 and 22
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Days
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Vibostolimab + Pembrolizumab After Crossover | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide
Number analyzed (Participants) | 48 | 230 | 0 | 0 | 0 | 0
Days
  Vibostolimab 2.10 mg Cycle 1: number analyzed (Participants) | 3 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 2.10 mg Cycle 1 | 3.82 [0.752 to 19.4] | NA [NA to NA] — Insufficient timepoints available to calculate |  |  |  |
  Vibostolimab 7.00 mg Cycle 1: number analyzed (Participants) | 3 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 7.00 mg Cycle 1 | 4.04 [1.46 to 11.2] | NA [NA to NA] — Insufficient timepoints available to calculate |  |  |  |
  Vibostolimab 7.00 mg Cycle 4: number analyzed (Participants) | 3 | 1 | 0 | 0 | 0 | 0
  Vibostolimab 7.00 mg Cycle 4 | 3.54 [1.44 to 8.52] | NA [NA to NA] — Insufficient timepoints available to determine t1/2 |  |  |  |
  Vibostolimab 21.0 mg Cycle 1: number analyzed (Participants) | 3 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 21.0 mg Cycle 1 | 7.19 [4.53 to 11.4] | 7.11 [4.10 to 12.3] |  |  |  |
  Vibostolimab 21.0 mg Cycle 4: number analyzed (Participants) | 1 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 21.0 mg Cycle 4 | NA [NA to NA] — Insufficient timepoints available to determine t1/2 | 11.0 [7.21 to 16.7] |  |  |  |
  Vibostolimab 70.0 mg Cycle 1: number analyzed (Participants) | 4 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 70.0 mg Cycle 1 | 5.45 [1.05 to 28.3] | 6.55 [2.68 to 16.0] |  |  |  |
  Vibostolimab 200 mg Cycle 1 | 7.58 [6.35 to 9.05] | 7.38 [6.92 to 7.87] |  |  |  |
  Vibostolimab 200 mg Cycle 4: number analyzed (Participants) | 18 | 124 | 0 | 0 | 0 | 0
  Vibostolimab 200 mg Cycle 4 | 11.6 [8.31 to 16.1] | 10.5 [9.71 to 11.5] |  |  |  |
  Vibostolimab 700 mg Cycle 1: number analyzed (Participants) | 7 | 49 | 0 | 0 | 0 | 0
  Vibostolimab 700 mg Cycle 1 | 6.04 [3.35 to 10.9] | 8.42 [7.44 to 9.53] |  |  |  |
  Vibostolimab 700 mg Cycle 4: number analyzed (Participants) | 4 | 26 | 0 | 0 | 0 | 0
  Vibostolimab 700 mg Cycle 4 | 8.39 [2.26 to 31.1] | 10.7 [9.16 to 12.6] |  |  |  |

20. Secondary Outcome: t1/2 of Plasma Vibostolimab Following Treatment With 200 mg Vibostolimab Combined With Various Other Treatments
Description: Blood samples were collected from participants during cycle 1 and cycle 4 of treatment (Cycle length is 21 days) following treatment with 200 mg vibostolimab in order to determine thet1/2 of plasma vibostolimab,
Time Frame: Cycle 1, Cycle 4: Day 1 pre-dose, 0.5 and 2 hours post-dose; once daily on Days 2, 3, 5, 8, 15 and 22
Population: Participants who complied with the protocol sufficiently to ensure that the data they generated will be likely to exhibit the effects of treatment, according to the underlying scientific model. Compliance covers such considerations as exposure to treatment, availability of measurements, and absence of major protocol violations. Cycle 4 for participants treated with etoposide was not analyzed due to insufficient time points available to determine t1/2.
Measure: Geometric Mean (95% Confidence Interval); unit: Days
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Vibostolimab + Pembrolizumab After Crossover | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide
Number analyzed (Participants) | 0 | 230 | 0 | 60 | 10 | 38
Days
  200 mg vibostolimab Cycle 1 |  | 7.38 [6.92 to 7.87] |  | 9.09 [8.33 to 9.91] | 5.38 [3.31 to 8.73] | NA [NA to NA] — Insufficient concentration time points available to calculate t1/2
  200 mg vibostolimab Cycle 4: number analyzed (Participants) | 0 | 124 | 0 | 19 | 8 | 0
  200 mg vibostolimab Cycle 4 |  | 10.5 [9.71 to 11.5] |  | NA [NA to NA] — Insufficient concentration time points available to calculate t1/2 | 10.5 [6.68 to 16.6] |

21. Secondary Outcome: t1/2 of Plasma Pembrolizumab Following Treatment With Increasing Amounts of Vibostolimab With 200 mg Pembrolizumab
Description: Blood samples were collected from participants during cycle 1 and cycle 4 of treatment (Cycle length is 21 days) in order to determine the t1/2 of plasma vibostolimab, Only results from participants treated with increasing amounts of vibostolimab combined with 200 mg pembrolizumab are presented; whereas other treatment groups were not analyzed.
Time Frame: Cycle 1, Cycle 4: Day 1 pre-dose, 0.5 and 2 hours post-dose; once daily on Days 2, 3, 5, 8, 15 and 22
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Days
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Vibostolimab + Pembrolizumab After Crossover | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide
Number analyzed (Participants) | 0 | 229 | 0 | 0 | 0 | 0
Days
  Vibostolimab 2.10 mg Cycle 1: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 2.10 mg Cycle 1 |  | 19.6 [12.0 to 31.9] |  |  |  |
  Vibostolimab 7.00 mg Cycle 1: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 7.00 mg Cycle 1 |  | 20.1 [14.6 to 27.7] |  |  |  |
  Vibostolimab 7.00 mg Cycle 4: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Vibostolimab 7.00 mg Cycle 4 |  | NA [NA to NA] — Due to insufficient data, results were not analyzed |  |  |  |
  Vibostolimab 21.0 mg Cycle 1: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 21.0 mg Cycle 1 |  | 8.84 [6.29 to 12.4] |  |  |  |
  Vibostolimab 21.0 mg Cycle 4: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 21.0 mg Cycle 4 |  | 18.6 [13.0 to 26.8] |  |  |  |
  Vibostolimab 70.0 mg Cycle 1: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0 | 0
  Vibostolimab 70.0 mg Cycle 1 |  | 13.1 [10.3 to 16.6] |  |  |  |
  Vibostolimab 200 mg Cycle 1 |  | 11.2 [10.6 to 11.8] |  |  |  |
  Vibostolimab 200 mg Cycle 4: number analyzed (Participants) | 0 | 124 | 0 | 0 | 0 | 0
  Vibostolimab 200 mg Cycle 4 |  | 14.3 [13.2 to 15.5] |  |  |  |
  Vibostolimab 700 mg Cycle 1: number analyzed (Participants) | 0 | 49 | 0 | 0 | 0 | 0
  Vibostolimab 700 mg Cycle 1 |  | 11.0 [9.95 to 12.2] |  |  |  |
  Vibostolimab 700 mg Cycle 4: number analyzed (Participants) | 0 | 26 | 0 | 0 | 0 | 0
  Vibostolimab 700 mg Cycle 4 |  | 16.1 [13.6 to 19.1] |  |  |  |

22. Secondary Outcome: t1/2 of Plasma Pembrolizumab Following Treatment With 200 mg Vibostolimab and 200 mg Pembrolizumab Combined With Various Other Treatments
Description: Blood samples were collected from participants during cycle 1 and cycle 4 of treatment (Cycle length is 21 days) following treatment with 200 mg vibostolimab and 200 mg pembrolizumab in order to determine the t1/2 of plasma pembrolizumab.
Time Frame: Cycle 1, Cycle 4: Day 1 pre-dose, 0.5 and 2 hours post-dose; once daily on Days 2, 3, 5, 8, 15 and 22
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: Days
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Vibostolimab + Pembrolizumab After Crossover | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide
Number analyzed (Participants) | 0 | 229 | 0 | 60 | 10 | 39
Days
  Cycle 1 |  | 11.2 [10.6 to 11.8] |  | 12.4 [11.1 to 13.8] | 16.6 [12.6 to 21.9] | NA [NA to NA] — Insufficient concentration time points available to calculate t1/2
  Cycle 4: number analyzed (Participants) | 0 | 124 | 0 | 19 | 8 | 0
  Cycle 4 |  | 14.3 [13.2 to 15.5] |  | NA [NA to NA] — Insufficient concentration time points available to calculate t1/2 | 17.7 [14.8 to 21.3] |

23. Secondary Outcome: Number of Participants Experiencing a Dose-Limiting Toxicity (DLT) at the End of Cycle 1
Description: A DLT is defined as an event with toxicity including the type, severity, time of onset, time of resolution, and the probable association with study treatment that are not due to pre-existing conditions as defined by CTCAE 4.0
Time Frame: At the end of Cycle 1 (up to 21 days)
Population: The population analyzed was treated participants. Per protocol, participants were assigned to a treatment group based on their unique combination of interventions. Hence for dose escalation, participants were assigned. to either monotherapy or sequential treatment groups rather than by dosage levels.
Measure: Count of Participants; unit: Participants
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Vibostolimab + Pembrolizumab After Crossover | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide
Number analyzed (Participants) | 68 | 293 | 25 | 60 | 10 | 40
Participants | 0 | 0 | 0 | 0 | 1 | 0

24. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) up to 24 Months
Description: A DLT is defined as an event with toxicity including the type, severity, time of onset, time of resolution, and the probable association with study treatment that are not due to pre-existing conditions as defined by the Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE4.0).
Time Frame: Up to 24 Months
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Vibostolimab + Pembrolizumab After Crossover | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide
Number analyzed (Participants) | 68 | 293 | 25 | 60 | 10 | 40
Participants | 0 | 0 | 0 | 0 | 1 | 0

25. Primary Outcome: Number of Participants Who Experienced At Least One Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol specified procedure, whether or not considered related to the medicinal product or protocol specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an adverse event.
Time Frame: Up to 28 Months
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Vibostolimab + Pembrolizumab After Crossover | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide
Number analyzed (Participants) | 68 | 293 | 25 | 60 | 10 | 40
Participants | 67 | 284 | 24 | 60 | 10 | 40

26. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: as for outcome 25
Time Frame: Up to 24 Months
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Vibostolimab + Pembrolizumab After Crossover | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide
Number analyzed (Participants) | 68 | 293 | 25 | 60 | 10 | 40
Participants | 2 | 30 | 1 | 4 | 1 | 3

27. Secondary Outcome: Rate of Progression Free Survival (PFS) Per RECIST 1.1 at 6 Months
Description: The progression free survival (PFS) rate is the percentage of participants who achieve PFS as estimated by the Kaplan-Meier method. PFS is the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first using RECIST, version 1.1 as assessed by investigator review. PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. Rate of PFS was planned and therefore only reported for participants treated with vibostolimab in combination with pembrolizumab, carboplatin or cisplatin, and etoposide. Other treatment groups were not analyzed.
Time Frame: 6 months
Population: Participants with a baseline scan with measurable disease by investigator assessment who were administered a dose of study treatment regardless of dose level. Only participants treated with vibostolimab in combination with pembrolizumab, carboplatin or cisplatin, and etoposide were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Vibostolimab + Pembrolizumab After Crossover | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Vibostolimab +Pembrolizumab+Pemetrexed+Carboplatin | Vibostolimab+Pembrolizumab+Carboplatin OR Cisplatin+Etoposide
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 40
Percentage of participants |  |  |  |  |  | 35.0 [20.8 to 49.6]

ADVERSE EVENTS:
Time Frame: All-cause mortality (ACM): from allocation up to a maximum of 28 months. Adverse events (AEs): from start of treatment up to a maximum of 28 months.
Description: The ACM population were allocated participants; the AE population were treated participants. Per protocol disease progression of cancer was not considered an AE unless related to study drug. Hence the following AE preferred terms not related to the drug were excluded: Neoplasm progression, Malignant neoplasm progression and Disease progression. As it was pre-specified to report adverse events irrespective of dose levels, treatment groups were instead based on their combination of interventions.
Groups:
- Part B: Vibostolimab + Pembrolizumab + Pemetrexed + Carboplatin: Participants received a 200 mg dose of vibostolimab in combination with 200 mg pembrolizumab, 500 mg/m^2 pemetrexed, and Area Under Curve (AUC) 5 mg/mL/min carboplatin on Day 1 of each 21-day infusion cycle for up to 4 cycles followed by maintenance therapy with a 200 mg dose of vibostolimab in combination with 200 mg pembrolizumab and 500 mg/m^2 pemetrexed on Day 1 of each 21-day infusion cycle for up to an additional 31 cycles.
- Part B: Vibostolimab + Pembrolizumab + Carboplatin or Cisplatin + Etoposide: Participants received 200 mg vibostolimab in combination with 200 mg pembrolizumab, plus the investigator's choice of Area Under Curve (AUC) 5 mg/mL/min carboplatin OR 75 mg/m^2 cisplatin on Day 1 of each 21-day cycle plus 100 mg/m^2/day etoposide on Days 1-3 of each 21-day cycle for up to 4 cycles. Maintenance therapy with 200 mg vibostolimab in combination with 200 mg pembrolizumab on Day 1 of each 21-day cycle will continue for up to an additional 31 cycles. A participant will be allowed to switch from cisplatin to carboplatin in the event of an adverse event (AE), ineligibility for further cisplatin therapy, and/or the investigator considers switching to carboplatin to be in the best interest of the participant.
Arm/Group | Vibostolimab | Vibostolimab + Pembrolizumab | Vibostolimab + Pembrolizumab After Crossover | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) | Part B: Vibostolimab + Pembrolizumab + Pemetrexed + Carboplatin | Part B: Vibostolimab + Pembrolizumab + Carboplatin or Cisplatin + Etoposide
All-Cause Mortality (participants affected / at risk) | 60/68 | 243/295 | 22/25 | 39/60 | 11/11 | 33/40
Serious Adverse Events (participants affected / at risk) | 18/68 | 99/293 | 7/25 | 26/60 | 5/10 | 13/40
Other Adverse Events (participants affected / at risk) | 64/68 | 274/293 | 23/25 | 60/60 | 10/10 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vibostolimab (N=68) | Vibostolimab + Pembrolizumab (N=293) | Vibostolimab + Pembrolizumab After Crossover (N=25) | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) (N=60) | Part B: Vibostolimab + Pembrolizumab + Pemetrexed + Carboplatin (N=10) | Part B: Vibostolimab + Pembrolizumab + Carboplatin or Cisplatin + Etoposide (N=40)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Addison's disease (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erosive duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 5 (5) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Malignant ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
H1N1 influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 10 (12) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma prolapse (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular insufficiency (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 5 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurogenic bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (6) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vibostolimab (N=68) | Vibostolimab + Pembrolizumab (N=293) | Vibostolimab + Pembrolizumab After Crossover (N=25) | Pembrolizumab/Vibostolimab Coformulation (MK-7684A) (N=60) | Part B: Vibostolimab + Pembrolizumab + Pemetrexed + Carboplatin (N=10) | Part B: Vibostolimab + Pembrolizumab + Carboplatin or Cisplatin + Etoposide (N=40)
Anaemia (Blood and lymphatic system disorders) | 17 (19) | 65 (85) | 4 (5) | 20 (39) | 4 (5) | 11 (12)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 14 (14) | 0 (0) | 3 (4) | 0 (0) | 4 (4)
Hypothyroidism (Endocrine disorders) | 1 (1) | 23 (23) | 0 (0) | 5 (5) | 0 (0) | 4 (4)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 5 (5) | 1 (1) | 6 (8) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 8 (9) | 41 (43) | 0 (0) | 6 (7) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 18 (18) | 2 (2) | 5 (5) | 1 (1) | 2 (2)
Ascites (Gastrointestinal disorders) | 4 (4) | 8 (9) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 6 (7) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 9 (9) | 43 (45) | 5 (5) | 9 (10) | 3 (3) | 12 (16)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 41 (56) | 3 (3) | 13 (14) | 3 (5) | 7 (12)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 10 (10) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 13 (14) | 70 (87) | 4 (4) | 19 (24) | 2 (2) | 14 (19)
Oral pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 11 (13) | 0 (0) | 2 (2) | 2 (2) | 5 (5)
Vomiting (Gastrointestinal disorders) | 7 (7) | 39 (51) | 2 (2) | 11 (15) | 1 (1) | 2 (4)
Asthenia (General disorders) | 3 (3) | 18 (18) | 1 (1) | 5 (5) | 2 (2) | 1 (1)
Chills (General disorders) | 3 (3) | 23 (24) | 0 (0) | 8 (8) | 0 (0) | 1 (2)
Fatigue (General disorders) | 21 (25) | 79 (89) | 7 (9) | 21 (24) | 5 (5) | 8 (9)
Gait disturbance (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Infusion site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 6 (6) | 25 (37) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Pain (General disorders) | 2 (2) | 5 (6) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (5) | 57 (84) | 2 (2) | 7 (8) | 1 (1) | 7 (7)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 5 (7) | 0 (0) | 1 (1) | 0 (0) | 4 (6)
Pneumonia (Infections and infestations) | 3 (3) | 7 (8) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Urinary tract infection (Infections and infestations) | 3 (3) | 18 (25) | 1 (1) | 3 (4) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 6 (6) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (3) | 15 (18) | 0 (0) | 1 (1) | 1 (1) | 7 (10)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (4) | 20 (24) | 0 (0) | 14 (23) | 1 (1) | 8 (9)
Amylase increased (Investigations) | 0 (0) | 17 (25) | 0 (0) | 9 (15) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 27 (33) | 1 (1) | 14 (22) | 1 (1) | 5 (5)
Bilirubin conjugated increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 5 (10) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 15 (16) | 1 (1) | 9 (11) | 0 (0) | 3 (4)
Blood bilirubin increased (Investigations) | 2 (2) | 9 (11) | 1 (2) | 6 (12) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 6 (12) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 7 (17) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 13 (13) | 2 (2) | 7 (10) | 0 (0) | 3 (5)
Lipase increased (Investigations) | 3 (3) | 24 (33) | 3 (3) | 13 (24) | 1 (1) | 3 (3)
Lymphocyte count decreased (Investigations) | 1 (1) | 19 (29) | 1 (1) | 6 (12) | 0 (0) | 1 (5)
Neutrophil count decreased (Investigations) | 1 (1) | 7 (9) | 1 (2) | 6 (9) | 0 (0) | 22 (45)
Platelet count decreased (Investigations) | 0 (0) | 5 (7) | 0 (0) | 6 (6) | 0 (0) | 10 (14)
Weight decreased (Investigations) | 1 (1) | 17 (17) | 1 (1) | 8 (10) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 10 (18) | 0 (0) | 12 (21)
Decreased appetite (Metabolism and nutrition disorders) | 16 (17) | 40 (44) | 4 (4) | 15 (15) | 3 (3) | 12 (13)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 10 (11) | 0 (0) | 2 (2) | 4 (4) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (4) | 1 (1) | 12 (41) | 0 (0) | 1 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (4) | 27 (47) | 1 (1) | 14 (18) | 0 (0) | 2 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (6) | 1 (2) | 7 (10) | 1 (1) | 2 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 22 (28) | 1 (1) | 13 (23) | 1 (1) | 1 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 11 (18) | 1 (1) | 4 (5) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 29 (43) | 1 (1) | 14 (18) | 2 (2) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (13) | 36 (46) | 3 (3) | 4 (5) | 2 (2) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 34 (35) | 2 (2) | 6 (7) | 1 (1) | 7 (8)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 14 (16) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 10 (12) | 1 (1) | 5 (5) | 1 (1) | 1 (1)
Neck mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 16 (21) | 2 (3) | 5 (6) | 2 (2) | 2 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 6 (6) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 7 (7) | 26 (26) | 1 (1) | 7 (9) | 1 (1) | 1 (1)
Dysaesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 9 (9) | 31 (34) | 1 (1) | 7 (9) | 2 (2) | 1 (1)
Nervous system disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 7 (7) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 8 (8) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 16 (18) | 0 (0) | 9 (10) | 3 (3) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 33 (33) | 0 (0) | 3 (3) | 2 (2) | 2 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 27 (30) | 2 (2) | 7 (8) | 2 (2) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (13) | 0 (0) | 7 (7) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 9 (10) | 0 (0) | 0 (0) | 2 (2) | 1 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Lichen planus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (12) | 72 (84) | 5 (5) | 15 (16) | 2 (2) | 16 (21)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 12 (15) | 64 (81) | 2 (3) | 16 (21) | 2 (3) | 15 (17)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (5) | 11 (13) | 0 (0) | 8 (8) | 2 (2) | 5 (7)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 15 (21) | 0 (0) | 6 (7) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 2 (2) | 14 (18) | 1 (1) | 5 (5) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/13/NCT02964013/Prot_SAP_000.pdf